CLINICAL TRIAL: NCT00150878
Title: Randomized Phase III Comparison of 12 Gy TBI and Cyclophosphamide 120 mg/kg With Fludarabine 120 mg/Sqm and 8 Gy TBI Before Allogeneic Transplantation in Patients With Acute Myeloid Leukemia in First Remission
Brief Title: Standard vs. Reduced-Intensity Conditioning in Patients With Acute Myeloid Leukemia in First Remission
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insurance coverage reached
Sponsor: University Hospital Carl Gustav Carus (Other)
Responsible Party: University Hospital Dresden
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9005-2003
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Reduced-intensity conditioning; Fludarabine; Acute myeloid Leukemia; Treatment-related mortality
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 12 Gy/Cyclophosphamide (Other): Standard intensity conditioning
  Interventions: Other: Conditioning therapy
- 8 Gy /Fludarabine (Experimental): Reduced-intensity conditioning
  Interventions: Other: Conditioning therapy

INTERVENTIONS:
Other: Conditioning therapy — Preparation before allogeneic transplantation

SUMMARY:
The primary goal of the study is to show that the treatment-related mortality of allogeneic hematopoietic stem cell transplantation an be significantly reduced by using a combination of 8 Gy total-body-irradiation and fludarabine in comparison to the conventional combination of 12 Gy TBI and 120 mg/kg Cyclophosphamide.

DETAILED DESCRIPTION:
Transplant-related deaths because of extramedullary toxicity and graft-versus host disease remain the major causes for treatment-failure in patients with AMl receiving allogeneic hematopoietic stem cell transplantation.

In phase II study, M . Stelljes and coworkers could show, that a reduced dose of total-body- irradiation and fludarabine can be safely used in patients with AML at various disease stages. The best results could be achieved in patients who had been in complete remission by the time of inclusion.

Therefore this prospective trial was initiated to compare the new conditioning regimen with the standard regimen of 12 Gy TBI/Cyclophosphamide 120 mg/kg in patients ith AML in first remission.

After having achieved complete remission, and giving informed consent, patients are stratified according to marrow cytogenetics, age and type of induction therapy and subsequently randomized to receive on of the mentioned conditioning therapies.

The primary end-point will be non-relapse mortality. The hypothesis would be, that the one-year mortality can be reduced from 25 to 15%. Given a power of 0.8 and a first-error of 5%, 252 patients will have to be randomized.

Secondary endpoints include:

3 year overall-and disease-free survival Rate of grade II-IV acute GvHD Rate of grade 3-4 extramedullary toxicity

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute myeloid leukemia in first remission
* Standard-or high-risk marrow cytogenetics
* HLA-matched related or unrelated donor available (in case of high-risk disease)
* Age 18 to 60
* Informed consent
* Consent of donor to donate peripheral blood stem cells
* sufficient liver function (elevation of transferases < 2.5 x upper limit)

Exclusion Criteria:

* AML with t(5;17)
* AML with t((8;21)
* clinically relevant heart failure (NYHA II-IV)
* Renal failure (creatinine > 200 µg/ml)
* Liver function failure (bilirubin > 3 mg/dl)
* Concomitant Neurological or psychiatric disease
* Contraindications to receive prescribed study medication
* HIV infection
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2003-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Treatment-related mortality at 12 months after transplantation | 12 months
  Proportion of patients dying without prior relapse

SECONDARY OUTCOMES:
Disease-free and Overall survival | 5 years
  Proportion of patients alive without relapse
Grade 3-4 extramedullary toxicity | 100 days
  Percentage of patients with grade II-IV acute GvHD

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Ehninger, MD, Study Director — Director of Med. Klink und Poliklinik I, Technical University Dresden
Locations (1):
- Medizinische Klinik und Poliklinik I, Dresden, Germany

REFERENCES:
- [Background] Stelljes M, Bornhauser M, Kroger M, Beyer J, Sauerland MC, Heinecke A, Berning B, Scheffold C, Silling G, Buchner T, Neubauer A, Fauser AA, Ehninger G, Berdel WE, Kienast J; Cooperative German Transplant Study Group. Conditioning with 8-Gy total body irradiation and fludarabine for allogeneic hematopoietic stem cell transplantation in acute myeloid leukemia. Blood. 2005 Nov 1;106(9):3314-21. doi: 10.1182/blood-2005-04-1377. Epub 2005 Jul 14. PMID 16020510
- [Derived] Fasslrinner F, Schetelig J, Burchert A, Kramer M, Trenschel R, Hegenbart U, Stadler M, Schafer-Eckart K, Batzel M, Eich H, Stuschke M, Engenhart-Cabillic R, Krause M, Dreger P, Neubauer A, Ehninger G, Beelen D, Berdel WE, Siepmann T, Stelljes M, Bornhauser M. Long-term efficacy of reduced-intensity versus myeloablative conditioning before allogeneic haemopoietic cell transplantation in patients with acute myeloid leukaemia in first complete remission: retrospective follow-up of an open-label, randomised phase 3 trial. Lancet Haematol. 2018 Apr;5(4):e161-e169. doi: 10.1016/S2352-3026(18)30022-X. Epub 2018 Mar 14. PMID 29550384
- [Derived] Bornhauser M, Kienast J, Trenschel R, Burchert A, Hegenbart U, Stadler M, Baurmann H, Schafer-Eckart K, Holler E, Kroger N, Schmid C, Einsele H, Kiehl MG, Hiddemann W, Schwerdtfeger R, Buchholz S, Dreger P, Neubauer A, Berdel WE, Ehninger G, Beelen DW, Schetelig J, Stelljes M. Reduced-intensity conditioning versus standard conditioning before allogeneic haemopoietic cell transplantation in patients with acute myeloid leukaemia in first complete remission: a prospective, open-label randomised phase 3 trial. Lancet Oncol. 2012 Oct;13(10):1035-44. doi: 10.1016/S1470-2045(12)70349-2. Epub 2012 Sep 7. PMID 22959335
- See also: Central Leukemia Study Group — http://www.kompetenznetz-leukaemie.de/